CLINICAL TRIAL: NCT05634291
Title: Effects of the Nottingham Arthritis App for Arthritis Pain
Brief Title: Effects of the Nottingham Augmented Reality (AR) App for Arthritis Hand Joint Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VRx Medical Inc (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); San Diego Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H210106
Record Dates: First submitted 2022-11-21; First posted 2022-12-02 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-02

CONDITIONS: Chronic Pain; Arthritis Hand; Opioid Use
Keywords: Augmented Reality; Smartphone application; Digital Therapeutic
MeSH Terms: conditions — Chronic Pain | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard of Care followed by AR digital treatment (Experimental): Standard of care period without active intervention followed by Digital treatment with active intervention
  Interventions: Other: Standard of care; Device: Nottingham AR smartphone app with active intervention

INTERVENTIONS:
Other: Standard of care — Standard of care as prescribed by healthcare provider.
Device: Nottingham AR smartphone app with active intervention — AR software treatment delivered by smartphone app and developed by VRx Medical (VRx) using established principles of illusion therapies (e.g. mirror therapy) for pain management.

SUMMARY:
The aim of this run-in design, feasibility study is to assess outcomes (including opioid-use, pain intensity, emotional function, and general physical function) for an augmented reality illusion therapy in participants with chronic hand joint pain due to arthritis.

DETAILED DESCRIPTION:
This is a run-in design, feasibility study that uses the enrolled participants as their own control. After consenting to join the study, for the first 30 days, participants will be on their current Standard of Care (SoC). Then, for the next 30 days, the same group of participants will use the Nottingham digital treatment daily. Pre- and Post-SoC and Treatment period measures of opioid use and pain, quality of life measures will be administered and measured. Additionally, for qualifying participants, Pre- and Post-treatment functional Magnetic Resonance Imaging (fMRI) scans will be performed to assess how Nottingham AR therapy affects neuroplastic changes in the supraspinal pain network associated with the therapy sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults ages 21-80
2. Clinical diagnosis of chronic hand pain from arthritis or as determined by study physician 3) Hand joint pain at a severity of 4 and above (on a 0 to 10 scale) daily

4) Use of prescribed opioids 5) English-speaking, literate, with stable residence 5) Able to operate a smartphone as evidenced by direct observation.

Exclusion Criteria:

1. Major medical illness that might confound effects of pain on function (e.g., advanced cardiac or pulmonary disease)
2. Current active alcohol or substance use disorder as evidenced from medical record
3. Currently active unstable psychiatric status in previous three months as measured by direct observation, patient self-report, or medical record
4. Moderate or severe cognitive impairment as demonstrated by medical diagnosis or clinical observation
5. fMRI exclusion only: Any factors that would prevent participation in fMRI

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
The Pain, Enjoyment of Life and General Activity scale (PEG) | Change from baseline to day 30
  PEG is a three-Item scale assessing pain intensity and interference. Scale is from 0 (no pain) to 10 (pain as bad as you can imagine).
Milligrams of Morphine Equivalent (MME) | Change from baseline to day 30
  MME is a standard measure of opioid use

SECONDARY OUTCOMES:
Resting State brain imaging data | Change from baseline to day 30
  fMRI compare pre- to post treatment - imaging data to show hyperactivities and enhanced functional connectivity in supraspinal regions associated with the affective aspect of pain perception.
Non-opioid pain medicine usage | Change from baseline to day 30
  Pain medicine usage will be tracked for dose and frequency.
Pain Disability Index (PDI) | Change from baseline to day 30
  PDI is a standard questionnaire designed to help patients measure the degree their daily lives are disrupted by chronic pain.
Patient Health Questionnaire (PHQ-9) | Change from baseline to day 30
  PHQ-9, a Quick Depression Assessment, is a reliable and valid measure of depression. severity

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rutledge, PhD, Principal Investigator — San Diego Veterans Healthcare System
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No